CLINICAL TRIAL: NCT00522821
Title: Treatment in Patients With Recurrent Infections and IgG Subclass Deficiency, and/or Deficient Anti-Polysaccharide Antibody Response
Brief Title: Treatment of Deficient Subclass or Anti-polysaccharide Antibody Response
Acronym: Subklasse
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IUWP2005.01
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-04

CONDITIONS: IgG Deficiency; Infections
Keywords: IgG subclass deficiency; Anti-polysaccharide deficiency; therapy; Immunoglobulins, Intravenous; co-trimoxazole
MeSH Terms: conditions — IgG Deficiency; Infections | interventions — Immunoglobulins, Intravenous; Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Antibiotics (Other): A: co-trimoxazole prophylactically for 12 months followed by intravenous immunoglobulin treatment for 12 months.
  Treatments will be separated by a washout period of 3 months during which co-trimoxazole will be given.
  Interventions: Drug: intravenous immunoglobulins; Drug: antibiotics
- intravenous immunoglobulins (Other): B: intravenous immunoglobulin treatment for 12 months followed by co-trimoxazole prophylactically for 12 months.
  Treatments will be separated by a washout period of 3 months during which co-trimoxazole will be given.
  Interventions: Drug: intravenous immunoglobulins; Drug: antibiotics

INTERVENTIONS:
Drug: intravenous immunoglobulins — * Adults: 600 mg/kg bodyweight every 3 weeks
  * Children: 800 mg/kg bodyweight every 3 week
  Other Names: Nanogam
Drug: antibiotics — * Children ≥5-12: If well tolerated, 4 mg trimethoprim and 20 mg sulfamethoxazole per kg bodyweight once daily, every day of the week (max160/800mg/day), combined with 5 mg folic acid.
  * Adults and children ≥12 years or ≥40 kg: If well tolerated, 160 mg trimethoprim and 800 mg sulfamethoxazole once daily, every day of the week combined with 5 mg folic acid.
  Other Names: co-trimoxazol; if not lorated: azitromycine

SUMMARY:
There is no consensus on the treatment of patients with recurrent infections and isolated immunoglobulin G (IgG)-subclass deficiency and/or selective antipolysaccharide antibody deficiency. Therefore, the Dutch Inter University Working Party will start a study in which the treatment with antibiotics is compared with intravenous immunoglobulin therapy with respect to clinical outcome measures in both children and adults with this disorder.

DETAILED DESCRIPTION:
There is no consensus on the treatment of patients with recurrent infections and isolated IgG-subclass deficiency and/or selective antipolysaccharide antibody deficiency. At present, there are no robust criteria to predict which patient will or will not respond adequately to antibiotic treatment or to IVIG. Furthermore, it is unknown whether IVIG treatment improves the quality of life in these patients. Therefore, the Dutch InterUniversity Working Party intends to start a study in this patient group. In this study, treatment for a year with antibiotics will be compared with a year intravenous immunoglobulin therapy with respect to clinical outcome measures in both children and adults with this disorder.

The patient will visit the clinic every 3 months during which laboratory tests and physiological measurements will be performed. Moreover the occurrence of infections and fever, the use of antibiotics, hospital admissions, and quality of life will be documented.

The study should result in a national harmonization in the treatment of this patient group. To this end, the results of the study will be used to compile a treatment protocol for this group of patients in the Netherlands and if applicable also in other countries worldwide.

ELIGIBILITY:
Inclusion Criteria:

* IgG subclass deficiency and/or (selective) antipolysaccharide antibody deficiency
* At least 2 physician documented infections before the start of the current treatment or in the last 6 months for newly diagnosed patients.
* Total serum IgG > 4 g/l
* ≥ 5 years of age
* Informed consent

Exclusion Criteria:

* Treatment with any other investigational drug within 7 days prior to study entry, or previous enrolment in this study
* Allergic reactions against human plasma/plasma products, or co-trimoxazole
* An ongoing progressive terminal disease
* Pregnancy or lactation
* History of (transient) cerebrovascular accident or coronary insufficiency
* Renal insufficiency (plasma creatinin > 115 µmol/L; or creatinin clearance <20 ml/min)
* An ongoing active disease causing general symptoms e.g. chronic active hepatitis or persistent enterovirus infection with ongoing systemic complaints
* Detectable anti-IgA antibodies
* Active systemic lupus erythematosus (SLE)
* Glucose-6-phosphate hydrogenase deficiency

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
the number, duration and type of infection (including use of antibiotics to treat infections), days of fever, hospital admissions and, if applicable, days absent from school or work due to infections. | 27 months

SECONDARY OUTCOMES:
Safety will be monitored by occurrence of adverse events, vital signs, and laboratory measurements. | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: J T van Dissel, PhD, MD, Principal Investigator — LUMC; T W Kuijpers, PhD, MD, Principal Investigator — AIDS Malignancy Consortium; E AM Sanders, PhD, MD, Principal Investigator — UMCU
Locations (9):
- Netherlands (9):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - AMC, Amsterdam
  - VU, Amsterdam
  - UMCG, Groningen
  - LUMC, Leiden
  - AZM, Maastricht
  - UMC St Radboud, Nijmegen
  - Erasmus MC, Rotterdam
  - UMCU, Utrecht